CLINICAL TRIAL: NCT05314257
Title: Role of Granisetron in Preventing Hypotension After Spinal Anesthesia With Levobupivacaine in Rheumatic Patients Undergoing Elective Cesarean Section: A Randomized Clinical Trial
Brief Title: Role of Granisetron in Preventing Hypotension After Spinal Anesthesia With Levobupivacaine in Rheumatic Patients Undergoing Elective Cesarean Section
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Granisetron
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Granisetron
MeSH Terms: interventions — Granisetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group G (Active Comparator): IV granisetron 1mg
  Interventions: Drug: Granisetron Hydrochloride
- Group C (Placebo Comparator): IV 5ml of 0.9% normal saline
  Interventions: Other: 0.9% normal saline

INTERVENTIONS:
Drug: Granisetron Hydrochloride — IV granisetron 1mg
  Other Names: granisetron
  Arms: Group G
Other: 0.9% normal saline — IV 5ml of 0.9% normal saline
  Other Names: normal saline
  Arms: Group C

SUMMARY:
Cardiac disease in pregnancy is a high-risk condition and a major cause of maternal mortality and morbidity. Although direct or immediate death due to cardiovascular disease is rare, it is an important indirect cause of maternal death worldwide, with an attributable rate of two deaths per 100,000 pregnancies. Cardiovascular physiological changes during pregnancy impose an additional load on the cardiovascular system of women with underlying heart disease which increases morbidity and mortality during pregnancy and at the time of delivery. Among cardiac diseases, Rheumatic Heart Disease is the commonest cardiac disease complicating pregnancy.

DETAILED DESCRIPTION:
The subarachnoid block is the most used anesthesia technique for conducting a cesarean section. The incidence of hypotension following this procedure is as high as 20-40% in pregnant patients. Similarly, bradycardia is also commonly associated with post-SAB, and the reported incidence is around 13%. Spinal anesthesia results in sympathetic block leading to a decrease in systemic vascular resistance and hypotension. Hypotension caused by subarachnoid block is physiologically compensated by an increase in heart rate. However, if vagus nerve-mediated Bezold-Jarisch reflex gets stimulated, then the cardiac autonomic balance gets shifted towards the parasympathetic nervous system leading to bradycardia, which further precipitates hypotension.

Levobupivacaine is a highly potent long-acting local anesthetic with a comparatively slow onset of action. Compared to bupivacaine, it has a lower tendency to block deactivated cardiac sodium and potassium channels with a more rapid rate of dissociation. It has reduced cardiac toxicity on overdose intravenous administration due to its faster protein binding rate. Plain levobupivacaine is isobaric to CSF. One of its advantages is that it has a more expectable spread. Several studies have revealed the reduced occurrence of various side effects (such as nausea, vomiting, bradycardia, and hypotension) when levobupivacaine compared with bupivacaine for spinal anesthesia used for cesarean delivery. It has been suggested to use 12.5-13.5mg levobupivacaine for effective spinal anesthesia for cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatic female patients in the childbearing period scheduled for elective cesarean sections

Exclusion Criteria:

* Patients with eclampsia and pre-eclampsia history,
* uncontrolled diabetes mellitus, morbid obesity,
* coagulation abnormalities,
* vertebral deformities, also patients who refused regional anesthesia,
* having contraindications to spinal anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
post-spinal hypotension, and bradycardia | 24 hours postoperative
  post-spinal hypotension, and bradycardia in rheumatic patients undergoing elective cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chatterjee A, Gudiwada B, Mahanty PR, Kumar H, Nag DS, Ganguly PK, Shukla R. Effectiveness of Granisetron in Prevention of Hypotension Following Spinal Anaesthesia in Patients Undergoing Elective Caesarean Section. Cureus. 2020 Dec 16;12(12):e12113. doi: 10.7759/cureus.12113. PMID 33489528
- [Background] Fakherpour A, Ghaem H, Fattahi Z, Zaree S. Maternal and anaesthesia-related risk factors and incidence of spinal anaesthesia-induced hypotension in elective caesarean section: A multinomial logistic regression. Indian J Anaesth. 2018 Jan;62(1):36-46. doi: 10.4103/ija.IJA_416_17. PMID 29416149
- [Background] Sharma B, Koirala E, Regmi S, Dhungana J, Neupane BK, Bhattarai S. Rheumatic Heart Disease among Pregnant Women with Cardiac Diseases in a Tertiary Care Center of Nepal: A Descriptive Cross-sectional Study. JNMA J Nepal Med Assoc. 2021 May 25;59(237):468-472. doi: 10.31729/jnma.6177. PMID 34508429